CLINICAL TRIAL: NCT00839085
Title: Effect of Ascorbic Acid and Grape Seed Extract "Vitis Vinifera L." in Oxidative Stress Induced by on Pump Coronary Artery by Pass Grafting Surgery
Brief Title: Comparison of Ascorbic Acid and Grape Seed Extract in Oxidative Stress Induced by on Pump Heart Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tabriz University (Other)
Responsible Party: Dr Naser Safaei, Cardiovascular Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 8710
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: CABG-Induced Oxidative Stress
Keywords: CABG; on pump; Grape seed extract; Vit C; Oxidative stress
MeSH Terms: interventions — Grape Seed Extract; Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): normal procedure of CABG
- 2: GSE (Active Comparator): 100 mg GSE every 6h /Po, starting one day before surgery (4 doses in 24h)
  Interventions: Drug: GSE
- 3: Vit C (Active Comparator): 25 mg/kg through pump
  Interventions: Drug: Vit C (Ascorbic Acid)

INTERVENTIONS:
Drug: GSE — grape seed extract (100 mg/6h), PO
  Other Names: Grape Seed Extract
  Arms: 2: GSE
Drug: Vit C (Ascorbic Acid) — Vit C 25 mg/ kg
  Other Names: Ascorbic Acid
  Arms: 3: Vit C

SUMMARY:
Study aimed to compare the effect of grape seed extract and ascorbic acid in oxidative stress induced by on pump coronary artery by pass grafting surgery.

DETAILED DESCRIPTION:
This study aimed to compare the effect of grape seed extract and ascorbic acid in oxidative stress induced by on pump coronary artery by pass grafting surgery.

There are three groups in the study. 75 candidate of coronary artery by pass grafting surgery were assigned random allocation on the groups (25 in each group).

1. Control
2. GSE (100 mg/6h - PO, 24h before surgery)
3. Vit C (25 mg/kg in pump circulation during surgery)

ELIGIBILITY:
Inclusion Criteria:

* Candidates for elective CABG surgery with pump for first time
* 3VD

Exclusion Criteria:

* High risk patients
* Those who need another heart surgery beside CABG
* Urgent patients
* Diabetics
* Ischemic time more than 120 min

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-11; Primary Completion 2009-01 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
LVEF | Before and after CABG

SECONDARY OUTCOMES:
Total Antioxidant Capacity (TAC) | Before ischemia, after ischemia, after reperfusion
MDA | Before, middle and after CABG
GTX | Before ischemia, after ischemia, after reperfusion
SOD | Before ischemia, after ischemia, after reperfusion

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Babaei, Pharm D, PhD, Principal Investigator — Drug Applied Research Center, Tabriz Univ Med Sci; Naser Safaei, MD, Surgeon, Study Chair — Tabriz Univ Med Sci; Masood Pezaeshkian, MD, Principal Investigator — Tabriz Univ Med Sci; Alireza Yaghobi, MD, Principal Investigator — Tabriz Univ Med Sci; Ahmad Reza Jodati, MD, Principal Investigator — Tabriz Univ Med Sci; Hossein Babaei, Pharm D, PhD, Study Director — Tabriz Univ Med Sci; Rasoul Azarfarin, MD, Principal Investigator — Tabriz Univ Med Sci; Mohammad Ali Sheikhalizadeh, CCP, Study Director — Tabriz Univ Med Sci
Locations (1):
- Cardiovascular Research Center, Tabriz, East Azerbaijan Province, Iran